CLINICAL TRIAL: NCT01311102
Title: Double Blind, Randomized, Prospective Trial of Impact of Pain Scores on Intrauterine Lidocaine vs Normal Saline Infusion Before IUD Placement.
Brief Title: The Impact of Pain Scores on Intrauterine Lidocaine Versus Normal Saline Infusion at the Time of IUD Placement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Women's Health Care Clinic, Torrance, California (Other)
Responsible Party: Principal Investigator, Anita Nelson, Medical Director, Women's Health Care Clinic, Torrance, California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13531-01
Record Dates: First submitted 2010-06-21; First posted 2011-03-09 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2013-12

CONDITIONS: Pain
Keywords: Pain score; IUD placement
MeSH Terms: conditions — Pain | interventions — Lidocaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2% Lidocaine liquid (Experimental): 1.33cc of 2% liquid lidocaine infused in endo cervix and endometrium
  Interventions: Drug: Lidocaine
- Normal Saline (Placebo Comparator): 1.33cc of normal saline infused in endo cervix and endometrium
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lidocaine — 1.33 cc 2% liquid lidocaine
  Other Names: Lidocaine Hydrochloride; Xylocaine
  Arms: 2% Lidocaine liquid
Drug: Normal Saline — 1.33cc normal saline
  Other Names: Sodium chloride
  Arms: Normal Saline

SUMMARY:
The study hypothesis is that infusion of 2% lidocaine at the time of IUD placement will reduce pain scores related to that procedure. In a double blinded randomized trial of 60 women receiving either normal saline or lidocaine infused through an endometrial aspirator, pain scores will be obtained for each step of the IUD placement procedure and for the total experience.

DETAILED DESCRIPTION:
IUDs are the most frequently used method of reversible birth control. The placement procedure is straightforward, but can cause the women cramping and pain. Every woman is advised to take Ibuprofen or acetaminophen prior to her appointment. Gentle techniques and distraction are used to minimize discomfort. However, some women still have measurable pain during and immediately after the procedure.

Investigators have shown that infusion of 5cc of a 2% concentration of liquid lidocaine into the inside of the uterus can reduce the pain that is associated with other procedures, such as biopsies done of the lining of the uterus. The investigators seek to determine if a similar infusion made before IUD placement may reduce pain. Because pain is a subjective complaint and because plastic tubing is being used to sound the uterus instead of the usual metal probe (a uterine sound), the investigators have included a placebo arm with saline infusion. All women will receive oral medication in advance of IUD placement, so no woman will be subject to placebo only.

Those women undergoing routine screening for IUD candidacy will be approached. Medical and social history and routine laboratory testing are to be done. The risks, benefits, and side effects of IUD placement will be explained. They will sign consent forms for the IUD from both the manufacturer and the clinic before evaluation for possible inclusion in this study. Informed consent for the study will be obtained either at that visit or on the day of the IUD placement. All the routine IUD placement steps will be done and she will rate the pain score. A standardized pain scale from 1-10, with 10 being the worst pain in the patient's lifetime, will be used here and at every point in the study. Depth of the uterus will be determined by introducing a plastic tubing into the woman's uterus. This tubing will either be filled with 1.3cc of normal saline or 2% lidocaine. The liquid will be infused at certain points within the cervix and uterus. She will again be asked to rate her pain score for that procedure. The tubing will be removed and the IUD will be placed. After the IUD is in the correct position, but before removal of the tenaculum, she will again be asked to rate her pain score for that procedure. After the IUD placement procedure is complete and the patient is dressed, she will be asked to assign an overall pain score. Pain scores between placebo and study drug used will be compared (mean, median and range). Fisher T tests will be performed to determine statistical significance with the p< 0.05 as a cutoff. Sub-analysis will be done comparing scores of which women who have never been pregnant to those who have. If possible, comparisons of pain scores will be made for women who have had vaginal deliveries compared to those who delivered by C-section. The risks to the patient for this study intervention are minimal.

ELIGIBILITY:
Inclusion Criteria:

* Women eligible for IUD insertion
* Willing to give consent

Exclusion Criteria:

* Allergy to lidocaine
* Contraindications to IUD use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita L Nelson, M.D., Principal Investigator — Women's Health Care Clinic
Locations (1):
- Women's Health Care Clinic, Torrance, California, United States

REFERENCES:
- [Background] Dogan E, Celiloglu M, Sarihan E, Demir A. Anesthetic effect of intrauterine lidocaine plus naproxen sodium in endometrial biopsy. Obstet Gynecol. 2004 Feb;103(2):347-51. doi: 10.1097/01.AOG.0000109519.74229.30. PMID 14754707
- [Background] Trolice MP, Fishburne C Jr, McGrady S. Anesthetic efficacy of intrauterine lidocaine for endometrial biopsy: a randomized double-masked trial. Obstet Gynecol. 2000 Mar;95(3):345-7. doi: 10.1016/s0029-7844(99)00557-8. PMID 10711541
- [Background] Gupta N, Ghosh B, Mittal S. Comparison of oral naproxen and intrauterine lignocaine instillation for pain relief during hysterosalpingography. Int J Gynaecol Obstet. 2008 Sep;102(3):284-6. doi: 10.1016/j.ijgo.2008.04.013. Epub 2008 Jul 7. PMID 18603250
- [Background] Lau WC, Tam WH, Lo WK, Yuen PM. A randomised double-blind placebo-controlled trial of transcervical intrauterine local anaesthesia in outpatient hysteroscopy. BJOG. 2000 May;107(5):610-3. doi: 10.1111/j.1471-0528.2000.tb13301.x. PMID 10826574
- [Background] Guney M, Oral B, Bayhan G, Mungan T. Intrauterine lidocaine infusion for pain relief during saline solution infusion sonohysterography: a randomized, controlled trial. J Minim Invasive Gynecol. 2007 May-Jun;14(3):304-10. doi: 10.1016/j.jmig.2007.02.007. PMID 17478360
- [Background] Edelman A, Nichols MD, Leclair C, Jensen JT. Four percent intrauterine lidocaine infusion for pain management in first-trimester abortions. Obstet Gynecol. 2006 Feb;107(2 Pt 1):269-75. doi: 10.1097/01.AOG.0000194204.71925.4a. PMID 16449111
- [Background] Hui SK, Lee L, Ong C, Yu V, Ho LC. Intrauterine lignocaine as an anaesthetic during endometrial sampling: a randomised double-blind controlled trial. BJOG. 2006 Jan;113(1):53-7. doi: 10.1111/j.1471-0528.2005.00812.x. PMID 16398772
- [Background] Edelman A, Nichols MD, Leclair C, Astley S, Shy K, Jensen JT. Intrauterine lidocaine infusion for pain management in first-trimester abortions. Obstet Gynecol. 2004 Jun;103(6):1267-72. doi: 10.1097/01.AOG.0000127981.53911.0e. PMID 15172863
- [Background] Frishman GN, Spencer PK, Weitzen S, Plosker S, Shafi F. The use of intrauterine lidocaine to minimize pain during hysterosalpingography: a randomized trial. Obstet Gynecol. 2004 Jun;103(6):1261-6. doi: 10.1097/01.AOG.0000127370.66704.f5. PMID 15172862
- [Background] Costello MF, Horrowitz S, Steigrad S, Saif N, Bennett M, Ekangaki A. Transcervical intrauterine topical local anesthetic at hysterosalpingography: a prospective, randomized, double-blind, placebo-controlled trial. Fertil Steril. 2002 Nov;78(5):1116-22. doi: 10.1016/s0015-0282(02)03362-9. PMID 12414003
- [Background] Guney M, Oral B, Mungan T. Efficacy of intrauterine lidocaine for removal of a "lost" intrauterine device: a randomized, controlled trial. Obstet Gynecol. 2006 Jul;108(1):119-23. doi: 10.1097/01.AOG.0000223201.42144.80. PMID 16816065
- [Derived] Nelson AL, Fong JK. Intrauterine infusion of lidocaine does not reduce pain scores during IUD insertion. Contraception. 2013 Jul;88(1):37-40. doi: 10.1016/j.contraception.2012.12.009. Epub 2013 Jan 2. PMID 23375352

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine: Lidocaine : 1.33 cc of 2% liquid lidocaine
- Normal Saline: Normal Saline : 1.33cc of normal saline
Period: Overall Study
Arm/Group | Lidocaine | Normal Saline
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pilot study using a population of convenience within study location.
Groups:
- Lidocaine: Lidocaine : 1.33cc of 2% liquid lidocaine
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Normal Saline | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years]
  Age Range | 32.05 (Not reported) [20 to 43] | 32.06 (Not reported) [19 to 46] | 32.055 (Not reported) [19 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores During Overall IUD Placement
Description: Pain score on 0-9 scale obtained just before the patient left the examination room; with 0 being "no pain" and 9 being "worst pain in life."
Time Frame: Before patient left the examination room at conclusion of procedure
Measure: Mean (Standard Deviation); unit: units on a scale of 0-9
Arm/Group | Lidocaine | Normal Saline
Number analyzed (Participants) | 20 | 20
units on a scale of 0-9 | 2.12 (2.32) [0 to 9] | 1.73 (1.49) [0 to 9]

2. Primary Outcome: Pain During Tenaculum Placement
Description: Pain score on 0-9 scale for tenaculum placement (without anesthesia); with 0 being "no pain" and 9 being "worst pain in life." Taken to adjust for different pain thresholds among subjects
Time Frame: Immediately following tenaculum placement
Measure: Mean (Standard Deviation); unit: units on a scale of 0-9
Arm/Group | Lidocaine | Normal Saline
Number analyzed (Participants) | 20 | 20
units on a scale of 0-9 | 2.20 (2.42) | 2.70 (2.03)

3. Primary Outcome: Pain Measurement During Liquid Infusion/Sounding
Description: After liquid infused into three parts of the endometrial cavity: in the lower one third, the middle, and at the top of the cavity. Pain was scored on a 0-9 scale; with 0 being "no pain" and 9 being "worst pain in life."
Time Frame: Recorded at the end of the infusion
Measure: Mean (Standard Deviation); unit: units on a scale of 0-9
Arm/Group | Lidocaine | Normal Saline
Number analyzed (Participants) | 20 | 20
units on a scale of 0-9 | 2.50 (3.09) | 3.39 (3.16)

4. Primary Outcome: Pain During IUD Placement
Description: IUD was inserted following the manufacturer's instructions, and a pain score was immediately obtained. Pain was scored on 0-9 scale; with 0 being "no pain" and 9 being "worst pain in life."
Time Frame: Immediately after IUD placement
Measure: Mean (Standard Deviation); unit: units on a scale of 0-9
Groups:
- Lidocaine: Lidocaine : 1.33cc of 2% liquid lidocaine infused in endo cervix and endometrium
- Normal Saline: Normal Saline : 1.33cc of normal saline infused in endo cervix and endometrium.
Arm/Group | Lidocaine | Normal Saline
Number analyzed (Participants) | 20 | 20
units on a scale of 0-9 | 2.95 (2.61) | 3.68 (2.71)

ADVERSE EVENTS:
Arm/Group | Lidocaine | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
This was a small pilot study, so may have missed small differences in pain score. Based on the results obtained, a sample size of 418 subjects would be needed to detect a statistically significant difference in the pain scores.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No